CLINICAL TRIAL: NCT02598934
Title: A Prospective Open-Label, Multicenter Study to Evaluate the Change in Bone Turnover Markers After Once Monthly Oral Ibandronate Therapy in Treatment Naive Postmenopausal Osteoporosis Patients
Brief Title: A Study of Ibandronate (Boniva) to Evaluate Bone Turnover Markers in Women With Treatment-Naive Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18057
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (2):
- Ibandronate Group 1 (Experimental): Participants will receive a 6-month regimen with oral ibandronate, 150 mg once monthly. Group 1 will receive a physician consultation after 4 months of treatment to review bone turnover test results.
  Interventions: Drug: Ibandronate
- Ibandronate Group 2 (Experimental): Participants will receive a 6-month regimen with oral ibandronate, 150 mg once monthly. Group 2 will not receive a physician consultation.
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Participants will receive oral ibandronate, 150 mg once weekly, for approximately 6 months.
  Other Names: Bonviva/Boniva

SUMMARY:
This study will evaluate whether an early positive response to once-monthly oral ibandronate in treatment-naive participants with postmenopausal osteoporosis is predictive of efficacy later in treatment. The anticipated time on study treatment is 6 months, and the target sample size is 360 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Women newly diagnosed with postmenopausal osteoporosis
* Naive to prior bisphosphonate therapy

Exclusion Criteria:

* Inability to stand or sit upright for at least 60 minutes
* Inability to swallow a tablet whole
* Hypersensitivity to any component of ibandronate
* Hormone (estrogen) replacement therapy within last 3 months, or will start on therapy within next 6 months
* Other osteoporosis drug within last 3 months
* Malignant disease diagnosed within previous 10 years, except resected basal cell cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2004-08; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (51):
- United States (49):
  - Montgomery, Alabama
  - Chandler, Arizona
  - Peoria, Arizona
  - Hot Springs, Arkansas
  - Pine Bluff, Arkansas
  - Anaheim, California
  - Beverly Hills, California
  - Carmichael, California
  - Wilmington, Delaware
  - DeLand, Florida
  - Miami, Florida
  - Palm Habor, Florida
  - Palm Springs, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Rome, Georgia
  - Morton Grove, Illinois
  - Indianapolis, Indiana
  - Waterloo, Iowa
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Reistertown, Maryland
  - Olive Branch, Mississippi
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Bloomfield, New Jersey
  - New York, New York
  - The Bronx, New York
  - Morehead City, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Doylestown, Pennsylvania
  - Langhorne, Pennsylvania
  - Philadelphia, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Morristown, Tennessee
  - Murfreesboro, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Texarkana, Texas
  - Richmond, Virginia
  - Tacoma, Washington
  - Madison, Wisconsin
- Puerto Rico (2):
  - Ponce
  - San Juan

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibandronate (Consult Group): Participants received ibandronate 150-milligram (mg) tablet once a month and a combination of calcium plus vitamin D supplement twice daily for 6 months, and received physician consultation on bone turnover marker (BTM) response.
- Ibandronate (Non-consult Group): Participants received ibandronate 150-mg tablet once a month and a combination of calcium plus vitamin D supplement twice daily for 6 months, and did not receive physician consultation on BTM response.
Period: Overall Study
Arm/Group | Ibandronate (Consult Group) | Ibandronate (Non-consult Group)
Started | 154 | 154
Completed | 135 | 132
Not Completed | 19 | 22
Not completed — Adverse Event | 11 | 13
Not completed — Failure to Return | 3 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Administrative | 2 | 1
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All enrolled participants who received at least 1 dose of study medication.
Groups:
- Ibandronate (Consult Group): Participants received ibandronate 150-mg tablet once a month and a combination of calcium plus vitamin D supplement twice daily for 6 months, and received physician consultation on BTM response.
- Total: Total of all reporting groups
Arm/Group | Ibandronate (Consult Group) | Ibandronate (Non-consult Group) | Total
Number analyzed (Participants) | 154 | 154 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9.94) | 64.9 (9.69) | 65.1 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 154 | 308
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Month 6 in Serum C-terminal Telopeptide of Type 1 Collagen (CTX)
Description: Serum CTX is a measure of bone resorption and is measured as nanograms per milliliter (ng/mL). Percent change from Baseline to Month 6 was calculated using Month 6 value minus baseline value divided by baseline value, and then multiplied by 100. Data for this outcome measure was reported for all participants combined (Consult group plus Non-consult group).
Time Frame: Baseline, Month 6
Population: ITT population observed cases: all participants of ITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Ibandronate (All Participants): Participants received ibandronate 150-mg tablet once a month and a combination of calcium plus vitamin D supplement twice daily for 6 months.
  Depending on the physician consultation on BTM response, participants were randomized into consult group and non-consult group.
Arm/Group | Ibandronate (All Participants)
Number analyzed (Participants) | 260
percent change | -55.26 (57.255)

2. Secondary Outcome: Percent Change From Baseline to Month 6 in Urine N-terminal Telopeptide of Type 1 Collagen (NTX)
Description: Urine NTX is a measure of bone resorption and is measured as millimoles bone collagen equivalents per millimoles creatinine. Percent change from baseline to Month 6 was calculated using Month 6 value minus baseline value divided by baseline value, and then multiplied by 100. Data for this outcome measure was reported for all participants combined (Consult group plus Non-consult group).
Time Frame: Baseline, Month 6
Population: ITT population observed cases: all participants of ITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate (All Participants)
Number analyzed (Participants) | 204
percent change | -45.98 (28.421)

3. Secondary Outcome: Percent Change From Baseline to Month 6 in Serum Procollagen Type 1 N-terminal Propeptide (P1NP)
Description: Serum P1NP is a measure of bone resorption and is measured as ng/mL. Percent change from baseline to Month 6 was calculated using Month 6 value minus Baseline value divided by baseline value, and then multiplied by 100. Data for this outcome measure was reported for all participants combined (Consult group plus Non-consult group).
Time Frame: Baseline, Month 6
Population: ITT population observed cases: all participants of ITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate (All Participants)
Number analyzed (Participants) | 235
percent change | -58.14 (25.334)

4. Secondary Outcome: Percent Change From Baseline to Month 6 in Serum Osteocalcin
Description: Serum osteocalcin is a measure of bone resorption and is measured as ng/mL. Percent change from baseline to Month 6 was calculated using Month 6 value minus baseline value divided by baseline value, and then multiplied by 100. Data for this outcome measure was reported for all participants combined (Consult group plus Non-consult group).
Time Frame: Baseline, Month 6
Population: ITT population observed cases: all participants of ITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate (All Participants)
Number analyzed (Participants) | 248
percent change | -41.51 (19.448)

5. Secondary Outcome: Percent Change From Baseline to Month 6 in Serum Bone-Specific Alkaline Phosphatase (BSAP)
Description: Serum BSAP is a measure of bone resorption and is measured as ng/mL. Percent change from baseline to Month 6 was calculated using Month 6 value minus baseline value divided by baseline value, and then multiplied by 100. Data for this outcome measure was reported for all participants combined (Consult group plus Non-consult group).
Time Frame: Baseline, Month 6
Population: ITT population observed cases: all participants of ITT population with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate (All Participants)
Number analyzed (Participants) | 253
percent change | -35.34 (17.386)

6. Secondary Outcome: Percentage of Participants Who Were "Very Confident" or "Confident" to Items on the Boniva Confidence Scale (BCS) at Month 6
Description: The BCS is designed to measure the participant's confidence level that Boniva (ibandronate) therapy is effective in treating osteoporosis and reducing the risk of fracture. Response options ranged on a 5-point scale from 'Not At All Confident' to 'Very Confident.' A Boniva confidence responder was defined as a participant who reported a response of 'confident' or 'very confident' on the 2 items in BCS. (1) ibandronate was effective in treating osteoporosis and (2) ibandronate reduces the risk of breaking a bone.
Time Frame: Month 6
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate (Consult Group) | Ibandronate (Non-consult Group)
Number analyzed (Participants) | 154 | 154
percentage of participants
  (1) Effective in treating osteoporosis | 68.8 | 51.9
  (2) Reduces risk of breaking bone | 64.9 | 50.0
  (1) or (2) | 72.1 | 55.2
  (1) and (2) | 61.7 | 46.8
Statistical Analysis 1: Comparison: Ibandronate (Consult Group) vs Ibandronate (Non-consult Group); Test type: Superiority or Other; p = 0.002, Chi-squared, Corrected — P-value between Consult group and Non-consult group for the item in the BCS: ibandronate was effective in treating osteoporosis; Difference in percentage of participants = 16.9, 95% CI 2-sided [6.1 to 27.7]
Statistical Analysis 2: Comparison: Ibandronate (Consult Group) vs Ibandronate (Non-consult Group); Test type: Superiority or Other; p = 0.009, Chi-squared, Corrected — P-value between Consult group and Non-consult group for the item in the BCS: ibandronate reduces risk of breaking bone; Difference in percentage of participants = 14.9, 95% CI 2-sided [4.0 to 25.8]
Statistical Analysis 3: Comparison: Ibandronate (Consult Group) vs Ibandronate (Non-consult Group); Test type: Superiority or Other; p = 0.001, Chi-squared, Corrected; P-value between Consult group and Non-consult group for items in BCS: ibandronate effective in treating osteoporosis or reduces risk of breaking bone; Difference in percentage of participants = 16.9, 95% CI 2-sided [6.3 to 27.5]
Statistical Analysis 4: Comparison: Ibandronate (Consult Group) vs Ibandronate (Non-consult Group); Test type: Superiority or Other; p = 0.010, Chi-squared, Corrected — P-value between Consult group and Non-consult group for items in BCS: ibandronate effective in treating osteoporosis and reduces risk of breaking bone; Difference in percentage of participants = 14.9, 95% CI 2-sided [3.9 to 25.9]

ADVERSE EVENTS:
Time Frame: AEs were recorded from baseline through Month 6 and in the follow-up period (15 days after the final Month 6 visit).
Description: Safety population: All participants who received at least 1 dose of study medication and had at least 1 post-baseline safety measurement. Safety data was reported for all participants combined (Consult group plus Non-consult group).
Arm/Group | Ibandronate (All Participants)
Serious Adverse Events (participants affected / at risk) | 17/308
Other Adverse Events (participants affected / at risk) | 76/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (All Participants) (N=308)
Arrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Melena (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (All Participants) (N=308)
Diarrhoea (Gastrointestinal disorders) | 26
Upper respiratory tract infection (Infections and infestations) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Back pain (Musculoskeletal and connective tissue disorders) | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the Overall Study. The sponsor may request that the confidential information be deleted and/or the publication to be postponed inorder to present the Sponsor's intellectual property rights.